CLINICAL TRIAL: NCT03798561
Title: A Phase 1, Randomized, Double-Blind, Vehicle-Controlled Ascending Doses Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ASN008 Topical Gel in Healthy Volunteers and Subjects With Atopic Dermatitis
Brief Title: Study to Evaluate ASN008 Topical Gel (TG)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASN008-101
Record Dates: First submitted 2019-01-04; First posted 2019-01-10 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2020-05

CONDITIONS: Dermatitis, Atopic; Pruritus; Dermatitis Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Intervention Model Description: Phase 1, multicenter, double-blind, vehicle-controlled, randomized ascending doses trial.
Who Masked: Participant, Investigator
Masking Description: Part A: Double blinded, with exception of unblinded dispensing pharmacist Part B: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 82 µg/cm2 ASN008 TG or Placebo (Experimental): PART A: ASN008 TG 82 µg/cm2 single application in 7 days or Placebo TG (6 subjects ASN008: 2 subjects placebo) (6:2)
  Interventions: Drug: ASN008 TG; Drug: Placebo TG
- 164 µg/cm2 ASN008 TG or Placebo (Experimental): PART A: ASN008 TG 164 µg/cm2 single application in 7 days or Placebo (6:2)
  Interventions: Drug: ASN008 TG; Drug: Placebo TG
- 328 µg/cm2 ASN008 TG or Placebo (Experimental): Part A: ASN008 TG 328 µg/cm2 single application in 7 days or Placebo (6:2)
  Interventions: Drug: ASN008 TG; Drug: Placebo TG
- 492 µg/cm2 ASN008 TG or Placebo (Experimental): Part A: ASN008 TG 492 µg/cm2 single application in 7 days or Placebo (6:2)
  Interventions: Drug: ASN008 TG; Drug: Placebo TG
- ASN008 TG TBD Cohort 1 or Placebo (Experimental): Part B: ASN008 TG Cohort 1 daily application for 15 days or Placebo (9 subjects ASN008: 3 subjects Placebo) (9:3)
  Interventions: Drug: ASN008 TG; Drug: Placebo TG
- ASN008 TG TBD Cohort 2 or Placebo (Experimental): Part B: ASN008 TG Cohort 2 daily application for 15 days or Placebo (9:3)
  Interventions: Drug: ASN008 TG; Drug: Placebo TG
- ASN008 TG TBD Cohort 3 or Placebo (Experimental): Part B: Placebo TG Cohort 3 daily application for 15 days or Placebo (9:3)
  Interventions: Drug: ASN008 TG; Drug: Placebo TG

INTERVENTIONS:
Drug: ASN008 TG — ASN008 TG
Drug: Placebo TG — Placebo TG

SUMMARY:
This is an ascending dose escalation study to test the safety, tolerability and preliminary efficacy of ASN008 TG in first-in-human subjects

DETAILED DESCRIPTION:
This is a two part, randomized, blinded, vehicle-controlled study to determine a safe and tolerable dose of ASN008 TG. Part A will asses a single ascending dose of ASN008 TG in cohorts of healthy volunteers, while Part B will assess multiple ascending doses of TG, to be determined (TBD) based on Part A safety and tolerability, in patients with mild-to-moderate dermatitis. Results from Part A and B will characterize safety, tolerability and pharmacokinetics. Part B patients will be assessed for changes in pruritus based on a numerical rating scale (NRS) of pruritus at baseline and on Day 15.

ELIGIBILITY:
Inclusion Criteria:

Part A - Healthy Volunteers:

* Written informed consent obtained prior to any required study-related procedure
* Healthy female or male subject aged 18 to 65
* Willing to use medically effective methods of birth control
* Females of reproductive potential must have a negative serum pregnancy test at screening and negative serum or urine pregnancy test prior to first study drug application on Day 1
* Non-smoker (no nicotine products for at least 6 months prior to screening)
* BMI ≥18.5 kg/m2 and ≤32.0 kg/m2 with minimum weight of 60 kg

Part B- Subjects with AD:

* Written informed consent obtained prior to any required study-related procedure
* Confirmed diagnosis of active atopic dermatitis (AD)
* History of AD for at least 6 months prior to Day 1 with an investigator global assessment ≥3 and body surface area covered with 1-10% AD
* Pruritus score (NRS)≥ 5 at screening and NRS ≥7 on Day 1

Exclusion Criteria:

Both Part A and Part B:

* Pregnant or breast-feeding women
* Skin disease that may interfere with study assessments
* Febrile illness within 6 days prior to Day 1, history of cancer within 5 years of Day 1, major surgery within 8 weeks prior to Day1, known immunodeficiencies, positive for hepatitis B or C or HIV infection
* Significant medical/surgical history or condition or current physical/laboratory/ECG/ vitals signs abnormality that might compromise the subject
* Corrected QT duration ≥450 milliseconds or other significant ECG abnormality
* Received marketed or investigational biological agent within 12 weeks prior to Day 1 or JAK inhibitor or nonbiological product or device within 4 weeks of Day 1 or within 8 weeks of Day 1 if investigational product used or any drug/ substance that is a strong inhibitor or inducer of CYP3A4 or CYP2D6
* Suspected hypersensitivity/allergy to lidocaine
* Significant drug or alcohol abuse or mental illness in 2 years prior to Day 1

Part A Only- Healthy Volunteers:

-Used medications or skin emollients within 2 weeks prior to Day 1 unless approved by investigator and sponsor

Part B Only - Subjects with AD:

* Has infected atopic dermatitis
* Used dupilumab 12 weeks prior to Day 1
* Used doxepin, hydroxyzine or diphenhydramine, urea containing topical products within 1 week prior to Day 1
* Used systemic antibiotics or topical medicated treatment or other systemic treatments that could affect AD 2 weeks prior to Day 1
* Received any UV-B phototherapy, excimer laser treatment or psoralen-UV-A treatment within 4 weeks prior to Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of ASN008 topical gel to define a maximum tolerated dose (Part A and B) | Part A: 14 days; Part B: 22 days
  Analyze incidence of treatment-emergent adverse events (TEAE)

SECONDARY OUTCOMES:
Calculate area under the plasma concentration versus time curve (Part A and B) | 7 days and 16 days
  A plot of the concentration of ASN008 in plasma over time
Calculate the Pharmacokinetic Half-life (Part A and B) | 7 days and 16 days
  Derive maximum blood plasma concentration of Time required for ASN008 concentration to decrease by 50%
Calculate the Pharmacokinetic maximum concentration (Part A and B) | 7 days and 16 days
  Maximum concentration of ASN008 achieved after dosing
Change from baseline in pruritus NRS in AD subjects (Part B) | 22 days
  Numeric Rating Scale ranging from 0 to 10; 0 indicates no itching; 10 indicates worst possible itching; Rating of pruritis based degree, duration, direction, disability, and distribution
Change from baseline in Eczema Area and Severity Score (EASI) in AD subjects (Part B) | 22 days
  Measurement of area and severity of atopic dermatitis based on composite score 0 to 72 encompassing degree of erythema, induration, excoriation and lichenification; each scored from 0 to 3 with 0 indicating none and 3 indicating severe
Change from baseline in Investigator Global Assessment Score in AD subjects (Part B) | 22 Days
  5 point morphological assessment of overall disease severity scored from 0 to 4 with 0 indicating clear (no inflammation) and 4 indicating severe (marked erythema)

CONTACTS AND LOCATIONS:
Overall Officials: Niranjan Rao, PhD, Study Director — Asana BioSciences
Locations (5):
- United States (4):
  - Certified Research Associates, Cortland, New York
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - Progressive Clinical Research, San Antonio, Texas
  - Spaulding Research Clinic, Inc, West Bend, Wisconsin
- Innovaderm Recherches Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramachandran R, Thompson SK, Malkmus S, Mieda T, Lin JH, Gupta S, Yaksh TL. Topical Application of ASN008, a Permanently Charged Sodium Channel Blocker, Shows Robust Efficacy, a Rapid Onset, and Long Duration of Action in a Mouse Model of Pruritus. J Pharmacol Exp Ther. 2020 Sep;374(3):521-528. doi: 10.1124/jpet.120.265074. Epub 2020 Jul 2. PMID 32616515